CLINICAL TRIAL: NCT07382700
Title: Metabolic Characteristics of Plasma OxPLs in STEMI Patients and Its Value Analysis in Predicting MACEs Risk After PCI Surgery.
Brief Title: Metabolic Characteristics of Plasma OxPLs in STEMI Patients.
Status: Enrolling by invitation | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Other Study IDs: 2025004A
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: STEMI - ST-segment Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: Healthy people
- CAD: Stable coronary heart disease patient
- STEMI-M: Male patients with ST segment elevation myocardial infarction
- STEMI-F: female patients with ST segment elevation myocardial infarction

SUMMARY:
The goal of this observational study is to investigate the structural composition and metabolic characteristics of OxPLs in STEMI patients. Explore OxPLs characteristic fingerprint biomarkers from different populations and analyze OxPLs fingerprint spectra. Based on the OxPLs fingerprint of STEMI patients, a machine learning classifier is used to establish an artificial intelligence assisted post PCI MACE risk prediction system, achieving the transformation of basic research into clinical application.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the diagnostic criteria for STEMI (refer to the "Diagnosis and Treatment Guidelines for Acute ST Segment Elevation Myocardial Infarction (2021)")
* Agree to perform direct PCI
* The onset time is less than 12 hours and successfully undergoing emergency PCI treatment
* After admission, all STEMI patients are routinely treated with antiplatelet aggregation, anticoagulation, lipid-lowering, and anti myocardial remodeling drugs.

Exclusion Criteria:

* Previous history of myocardial infarction
* Accompanied by other cardiovascular diseases, such as severe heart valve disease, severe heart failure, congenital heart disease, cardiomyopathy, etc
* Merge with severe infection
* Merge with severe anemia
* Merge with severe liver and kidney dysfunction
* Combined with malignant tumors
* Accompanied by a history of autoimmune or hematological diseases
* Recent history of severe trauma or surgery
* Patients with incomplete clinical data
* The patient does not agree to undergo data collection

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: STEMI patients admitted to our cardiovascular department for concurrent PCI surgery between January 2025 and December 2025.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China